CLINICAL TRIAL: NCT06024577
Title: Aherence to Different Exercise Interventions
Brief Title: Adherence to Different Exercise Interventions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Chair and Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-152
Record Dates: First submitted 2023-07-01; First posted 2023-09-06 (Actual); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Exercise Adherence
MeSH Terms: interventions — Walking

STUDY DESIGN:
Intervention Model Description: Randomized study to three arms: 1) walk intervention, 2) variety intervention, 3) progressive intervention
Who Masked: Outcomes Assessor
Masking Description: Research staff collecting data will be masked to intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Walking (Active Comparator): Participants prescribed 150 minutes/week of moderate to vigorous walking.
  Interventions: Behavioral: Walking
- Variety (Experimental): Participants prescribed 150 minutes/week of moderate to vigorous variety of exercise. Each week participants will be prescribed a single different exercise (variety) which will include cycling, walking/jogging, yoga/Pilates, and cross-training.
  Interventions: Behavioral: Variety
- Progressive (Experimental): Participants prescribed 150 minutes/week of moderate to vigorous exercise. The exercises include cycling, walking/jogging, yoga/Pilates, and cross-training, and each week another exercise will be added to the list of options for participants. Participants may choose from the list of exercise. They do not have to do them all, and they can do as much or little (none) of whatever they choose.
  Interventions: Behavioral: Progressive

INTERVENTIONS:
Behavioral: Walking — Prescribed 150 minutes per week of moderate to vigorous walking.
  Arms: Walking
Behavioral: Variety — Prescribed 150 minutes per week of moderate to vigorous variety of exercise. Each week participants are randomly asked to participate in cycling, walking/jogging, yoga/Pilates, or cross-training.
  Arms: Variety
Behavioral: Progressive — Prescribed 150 minutes per week of moderate to vigorous progressive variety of exercise. Each week participants are randomly asked to participate in cycling, walking/jogging, yoga/Pilates, or cross-training. Participants can choose which exercise they want to do, and can do as much or little as they want.
  Arms: Progressive

SUMMARY:
Only 50% of sedentary adults that start an exercise training program adhere to the program after 6 months. Exercise variety may improve adherence. The goal of this study is to examine different exercise interventions that include a variety of exercise on adherence.

DETAILED DESCRIPTION:
Regular exercise, in the form of walking 150 minutes per week, is widely regarded as having many health and fitness benefits. Despite these well-known benefits, adherence to exercise interventions is extremely low. When sedentary adults start an exercise training program only 50% adhere to the program and meet the national recommendations of 150 minutes per week. A possible explanation of the low adherence is that most adults only walk for exercise, and that providing a variety of exercise may increase adherence. Preliminary observational data show that a variety of exercise may increase weekly exercise expenditure compared to other interventions. The overall objective of this study is to investigate the feasibility, adherence, and acceptability of different exercise interventions including 1) walk intervention, 2) variety intervention, and 3) progressive intervention (see below for description).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* Sedentary (<1 hour per week of exercise)
* BMI 18.5 to 40 kg/m2

Exclusion Criteria:

* Adults with diagnosed cardiovascular, diabetes, renal, or any other metabolic disease determined by Health and Fitness History questionnaire.
* Any other disability, ailment, or physical characteristics that may hinder the ability to participate in regular exercise determined by Health and Fitness History questionnaire.
* Participating in other studies that would interfere with their ability to safely complete the exercise protocols.
* Pregnant or trying to become pregnant, and peri-menopausal or post-menopausal women.
* History of smoking within the last 6 months
* Any other vulnerable population (children <18, pregnant women, prisoners, etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender criteria are:
  * Cisgender man (non transgender)
  * Cisgender woman (non transgender)
  * Transgender man
  * Transgender woman
Enrollment: 60 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Adherence to exercise intervention | Change from baseline at 1-week, 2-weeks, 3-weeks, and 4-weeks
  Adherence is assessed as meeting or exceeding 150 minutes per week of moderate to vigorous exercise

SECONDARY OUTCOMES:
Acceptability of intervention | Acceptability at 4-weeks
  Participants will complete a survey on acceptability at the end of the exercise intervention
Body Weight | Change in body weight from baseline to 4-weeks
  Body weight will be measured at baseline and 4-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hagobian, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and documentation will be available under a data-sharing agreement. Information shared with outside collaborators will link data to two unique study identifiers (de-Identified) to maintain participant anonymity, and outside researchers and the community will not be allowed to have access to participant names and confidential information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Seven years after the date of the last participant completing the study.
Access Criteria: Contact PI and a date-sharing agreement will be created that provides for (1) a commitment to use the data for research purposes only; (2) a commitment to securing the data using appropriate computer technology (password protected and encrypted); (3) a commitment to destroying or returning the data after analyses are completed and (4) a commitment not to attempt to identify participants individually.
URL: http://healthresearch.calpoly.edu/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT06024577/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT06024577/ICF_001.pdf